CLINICAL TRIAL: NCT06257212
Title: Using Live Vaccines to Induce Beneficial Innate Immune Training and Reduce Systemic Inflammation in COPD Patients.
Brief Title: Live Vaccines and Innate Immune Training in COPD.
Acronym: COPD-LIVE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Josefin Eklöf (Other)
Responsible Party: Sponsor-Investigator, Josefin Eklöf, MD, PhD, Chronic Obstructive Pulmonary Disease Trial Network, Denmark
Organization: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: COPD-LIVE
Record Dates: First submitted 2024-02-06; First posted 2024-02-13 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Trained Innate Immunity; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — BCG Vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Intervention Model Description: Single-blinded 1:1:1 block randomized controlled trial (with varying block sizes of 3-6), stratified by sex.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCG vaccine (Active Comparator): Intradermal BCG vaccine (0.1 ml) + subcutaneous saline at inclusion and after 3 months.
  Interventions: Drug: BCG vaccine (Danish strain 1331)
- MMR vaccine (Active Comparator): Subcutaneous MMR vaccine (0.5ml) + intradermal saline at inclusion and after 3 months.
  Interventions: Drug: MMR Vaccine
- Placebo (Placebo Comparator): Subcutaneous saline + intradermal saline at inclusion and after 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCG vaccine (Danish strain 1331) — Intradermal BCG vaccine (0.1 ml) + subcutaneous saline at inclusion and after 3 months.
  Arms: BCG vaccine
Drug: MMR Vaccine — Subcutaneous MMR vaccine (0.5ml) + intradermal saline at inclusion and after 3 months.
  Arms: MMR vaccine
Drug: Placebo — Subcutaneous saline + intradermal saline at inclusion and after 3 months.
  Arms: Placebo

SUMMARY:
A randomized, single-blinded clinical pilot study to assess whether vaccination with live attenuated vaccines can induce trained immunity and cause beneficial changes in patients with COPD.

DETAILED DESCRIPTION:
Single-blinded 1:1:1 block randomized controlled trial (with varying block sizes of 3-6), stratified by sex. A total of 60 participants will be recruited and randomly assigned with 20 in each treatment arm. Separated by three months, the participants will receive two doses of one of the following three treatments:

1. MMR vaccine (M-M-R VaxPro)
2. BCG vaccine (Danish strain 1331)
3. Saline (placebo)

ELIGIBILITY:
Inclusion Criteria:

* Specialist verified and spirometry-confirmed COPD
* Age > 40 years.
* Negative HIV-test.
* Able to give informed consent.

Exclusion Criteria:

* Acute febrile illness.
* Known allergy to BCG or MMR vaccines or serious adverse effects at previous vaccination.
* Allergy to MMR vaccine components, neomycin, or egg proteins.
* Known prior, active, or latent infection with mycobacterium tuberculosis.
* Pregnancy or breastfeeding.
* Vaccination with a live vaccine within the last 4 weeks.
* Being severely immunocompromised (HIV-1 infection, organ- or bone marrow transplantation, chemotherapy, primary immune defect, anti-cytokine therapy, immunosuppressant treatment).
* Oral or intravenous corticosteroid at dose of ≥10 mg/day with duration over 3 months.
* Active solid or non-solid malignancy or lymphoma, excluding basal cell carcinoma within 2 years.
* Treatment with immunoglobulins within the last 3 months or expected treatment with immunoglobulins for the duration of the trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Innate immune training. | From inclusion to 4 months post-inclusion.
  Innate immune training, detected as fold-changes in cytokine production capacity of innate immune cells for cytokines such as IL-1β, IL-6, IL-10, TNF-α and IFN-γ, following pro-inflammatory stimulation from inclusion to 4 months post-inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik Stæhr S Jensen, MD,Phd, Principal Investigator — Herlev Gentofte Hospital
Locations (1):
- Department of Internal Medicine, Section of Respiratory Medicine, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided